CLINICAL TRIAL: NCT04979130
Title: A Randomized Parallel Comparison of Semaglutide Versus Placebo on Intestinal Barrier Function in Type 2 Diabetes Mellitus (SIB)
Brief Title: Comparing Semaglutide Versus Placebo on Intestinal Barrier Function in Type 2 Diabetes Mellitus (SIB)
Acronym: SIB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21-2774
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Chronic Inflammation; Intestinal Permeability
Keywords: T2D; Type 2 diabetes; Type 2 diabetes mellitus; obesity; intestinal permeability; chronic inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SC semaglutide (Experimental): Participants receive a once weekly, subcutaneous, Semaglutide injection for 16 weeks in addition to the participants background metformin monotherapy. The participants in this arm will begin at a 0.25 mg dose during the randomization visit, at week 4 this will be escalated to a 0.5 mg dose and at week 8 it will be escalated again to a 1.0 mg dose if tolerable by the participant. If the participant cannot tolerate the 0.25 mg dose at randomization or the 0.5 mg dose at week 4 they will be withdrawn from the study.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants in this arm will be given a once weekly, subcutaneous, placebo injection matching the Semaglutide experimental arm in addition to their background metformin monotherapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide 1.34 mg/mL solution for injection in 1.5 mL pre-filled PDS290 pen-injector provided by Novo Nordisk.
  Other Names: Ozempic; PDS290 pen-injector
  Arms: SC semaglutide
Drug: Placebo — Semaglutide placebo, solution for injection, 1.5 mL pre-filled PDS290 pen-injector provided by Novo Nordisk.
  Other Names: PDS290 pen-injector
  Arms: Placebo

SUMMARY:
This study plans to learn more about the effect of semaglutide once weekly on intestinal permeability in individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial, except for protocol described pre-screening activities, which require a separate informed consent.
2. Male or female, age above or equal to 18 years at the time of signing informed consent.
3. Diagnosed with type 2 diabetes mellitus on metformin monotherapy
4. Hemoglobin A1c <8.0% (<64 mmol/mol) on screening day
5. Body mass index (BMI) ≥28 kg/m2
6. Low-grade inflammation, defined as elevated high sensitivity C-reactive protein (hs- CRP >1.0 and ≤10 mg/L). Impaired intestinal barrier function results in activation of inflammatory pathway; therefore, excluding subjects with no evidence of inflammation (hs-CRP ≤ 1 mg/L) will help to enrich our study population. Similar threshold for hs-CRP as a marker of "residual inflammatory risk" (29) has been previously used as an independent predictor of future vascular events (26, 30).

Exclusion Criteria:

1. Known or suspected hypersensitivity to trial product or related products.
2. Female who is pregnant, breast-feeding or intends to become pregnant or is of child- bearing potential and not using a highly effective contraceptive method.
3. Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days before screening.
4. Any disorder, which in the investigator's opinion might jeopardize patient's safety or compliance with the protocol.
5. Any of the following: myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischemic attack (TIA) within the past 60 days prior to the day of screening.
6. Second anti-diabetic agent use within 3 months of screening.
7. Chronic kidney disease defined as eGFR < 30 mL/min/1.73 m2.
8. C-reactive protein (hs-CRP >10.0 mg/L) to eliminate patients with acute inflammatory process at the time of screening.
9. Any recent infection or antibiotic use within 3 weeks
10. Regular use (more than a week duration) of anti-inflammatory medication (steroid or NSAIDs) within 3 months of screening.
11. Regular use (more than a week duration) of any digestive health supplements, such as probiotics or prebiotics within 3 months screening.
12. Diagnosis of chronic intestinal inflammatory disease such as Crohn's disease, ulcerative colitis or irritable bowel syndrome.
13. Prior bariatric or bowel surgery
14. Heart failure presently classified as being in New York Heart Association (NYHA) Class IV.
15. Presence or history of malignant neoplasm within 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ is allowed.
16. Personal or family history of multiple endocrine neoplasia type 2 (MEN2) or medullary thyroid carcinoma (MTC).
17. History of chronic pancreatitis or history of acute pancreatitis within 6 months of screening.
18. Chronic consumption of > 2 alcoholic standard drinks per day as defined by:

    * 12 ounces of beer (5% alcohol content).
    * 8 ounces of malt liquor (7% alcohol content).
    * 5 ounces of wine (12% alcohol content).
    * 1.5 ounces or a "shot" of 80-proof (40% alcohol content) distilled spirits or liquor (e.g., gin, rum, vodka, whiskey).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Differences in lactulose mannitol ratio (LMR) test as a measure of intestinal permeability between treatment groups | Week 16 (visit 6)
  The ratio of lactulose to mannitol will be measured in urine collected within 6 hours after ingestion of dual sugar. This ratio predominantly reflects small intestine permeability.

SECONDARY OUTCOMES:
Differences between treatment groups in plasma LBP | Week 8 (visit 4), Week 16 (visit 6)
  Marker of intestinal permeability
Differences between treatment groups in Serum zonulin | Week 8 (visit 4), Week 16 (visit 6)
  Marker of intestinal permeability
Differences between treatment groups in Fecal Calprotectin | Week 8 (visit 4), Week 16 (visit 6)
  Marker of intestinal inflammation
Differences between treatment groups in plasma IL-6 | Week 8 (visit 4), Week 16 (visit 6)
  Marker of chronic inflammation
Differences between treatment groups in plasma IL-8 | Week 8 (visit 4), Week 16 (visit 6)
  Marker of chronic inflammation
Differences between treatment groups in plasma TNFα | Week 8 (visit 4), Week 16 (visit 6)
  Marker of chronic inflammation
Differences between treatment groups in plasma hs-CRP | Week 8 (visit 4), Week 16 (visit 6)
  Marker of chronic inflammation

OTHER OUTCOMES:
Exploratory: determine the effect of semaglutide as compared to placebo on intestinal microbiota in relation to changes in intestinal permeability and inflammatory markers | Visit 6 (week 16)
  Microbiome study

CONTACTS AND LOCATIONS:
Overall Officials: Neda Rasouli, MD, Principal Investigator — University of Colorado, Denver; Joseph Onyiah, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States